CLINICAL TRIAL: NCT06325072
Title: Set-up of a Platform for Personalized Diagnosis of Rare Kidney Diseases (NIKE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paola Romagnani, MD, Meyer Children's Hospital IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NIKE
Record Dates: First submitted 2024-02-29; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Patients selected based on the inclusion criteria will be evaluated by a multidisciplinary team of experts. All the selected patients will undergo genetic testing by clinical exome sequencing and in silico filtering for a panel of genes described as causing or in association with CKD. Identified variants will be classified according to the American College of Medical Genetics and Genomics (ACMG) guidelines. Reverse phenotyping will be performed according to the results of genetic testing. The results of the diagnostic work-up will be evaluated by a multi-disciplinary team of experts in order to establish conclusive diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pathogenic variants (Experimental): Variants fitting bioinformatic prioritization criteria for pathogenicity according to ACMG guidelines and the clinical phenotype, and variants already reported in the literature will be defined as pathogenic variants
  Interventions: Diagnostic Test: Conclusive genetic testing
- Potentially Pathogenic Variants (Experimental): Variants fitting bioinformatic prioritization criteria but apparently do not correlate with the clinical phenotype and have not been previously reported in the literature will be defined as potentially pathogenic variants
  Interventions: Diagnostic Test: Genotype-phenotype correlation for personalized diagnosis
- Variants of Unknown Significance (VUS) (Experimental): Variants fitting the phenotype but not fitting bioinformatic prioritization criteria will be defined as variants of uncertain clinical significance (VUS)
  Interventions: Diagnostic Test: Personalized study of variants of uncertain clinical significance (VUS) through functional studies on 3D organ-on-a-chip

INTERVENTIONS:
Diagnostic Test: Conclusive genetic testing — Patients will be referred for genetic counseling at the study coordinating center. This will lead to a conclusive genetic diagnosis.
  Arms: Pathogenic variants
Diagnostic Test: Genotype-phenotype correlation for personalized diagnosis — Patients and their family members will undergo a thorough clinical reassessment at the study coordinating center to identify diagnostic handles of the suspected disease based on the genetic test result (reverse phenotyping). The clinical reassessment could include the performance of additional clinical and instrumental tests, as well as other specialized consultations. This will lead to a conclusive genetic diagnosis in a substantial proportion of cases, cases, who will then be provided with genetic counselling.
  Arms: Potentially Pathogenic Variants
Diagnostic Test: Personalized study of variants of uncertain clinical significance (VUS) through functional studies on 3D organ-on-a-chip — The investigators will perform functional assessment trough urine derived Renal Progenitor Cells (u-RPC) to establish the role of variants in determining the clinical phenotype.
  Arms: Variants of Unknown Significance (VUS)

SUMMARY:
Chronic kidney disease (CKD) is a major health problem, with steadily increasing incidence and prevalence and the threat of a true "epidemic". Converging evidence suggests a high prevalence of genetic etiology in rare kidney diseases and the list of new disease-causing genes is constantly updated. Recent advances in next-generation sequencing (NGS) technologies have prompted a significant improvement in the diagnosis of rare kidney diseases. Notwithstanding this, NGS generates high numbers of information that need to be properly analysed by the joint efforts of geneticists, nephrologists and bioinformatics in order to integrate clinical and genetic information in a personalized manner. In addition, in selected cases, the contribution of researchers proves essential for the development of experimental models of the disease to study and understand the pathogenic features and propose a personalized therapeutic approach. Such an innovative, integrated diagnostic paradigm is currently available in few centers all over the world and cannot be easily translated in daily clinical practice.

The aim of the study is to set-up an integrated diagnostic algorithm to extend the newest personalized diagnostic and treatment strategies for rare kidney diseases to all patients in the Tuscany region, under 40 years of age with kidney disease. This algorithm will be based on a constant cross-talk between participating centers and a dedicated multidisciplinary team. Diagnostic and therapeutic performances will be validated at European level.

ELIGIBILITY:
Inclusion Criteria:

* family history of kidney disease and/or parental consanguinity;
* extra-renal involvement (e.g., sensorineural hearing loss);
* resistance to treatment (e.g., immunosuppressive);
* metabolic acidosis or metabolic alkalosis in the absence of renal failure;
* ultrasound detection of of at least 2 cystic lesions in each kidney or nephrocalcinosis;
* ultrasound detection of congenital abnormalities of the kidney and urinary tract (CAKUT) and CKD stage ≥ 2 according to KDIGO definition
* informed consent form.

Exclusion Criteria:

* age > 40
* refuse to participate to the study

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Validation of genetic diagnosis | From enrollment (genetic testing) until the date of returning of genetic testing results (up to 6 months)
  The investigators will assess the role of potentially pathogenic variants and variants of uncertain clinical significance (VUS) in determining a conclusive genetic diagnosis by patient reassessment (reverse phenotyping) or in vitro functional studies.
  In detail, after the results of ES, a multidisciplinary team will evaluate the results of sequencing and will eventually request additional investigations (e.g., laboratory or imaging tests, specific consultations, etc) to the patient and/or family member in order to look for previously undetected/overlooked signs of the genetic diseases suggested by ES (reverse phenotyping).
  In vitro functional studies on u-RPC will be requested in a subset of patients. The number of patients with a conclusive diagnosis obtained trough these strategies will contribute to the overall diagnostic rate of the workflow (number of conclusive genetic diagnosis/number of patients enrolled in the study).

SECONDARY OUTCOMES:
Identification of molecular pathways | From enrollment (genetic testing) until the last patient last visit, estimated up to 12 months
  The investigators aim to o identify molecular pathways that could represent potential therapeutic targets in a selection of patients carrying potentially pathogenic variants.
  To this goal, the investigators will perform single-cell RNA sequencing on kidney biopsy fragments of patients who have undergone a diagnostic kidney biopsy. After obtaining intracellular transcriptome of individual cells carrying the potentially pathogenic variants, the investigators will compare their RNA expression profile to the same type of cells obtained from non-mutated patients.
Explore the applicability of gene editing in rare kidney diseases | From enrollment (genetic testing) until the last patient last visit, estimated up to 12 months
  The investigators will explore the applicability of CRISPR/Cas9 gene editing in rare kidney diseases through u-RPCs obtained from patients carrying pathogenic mutations.
  In order to achieve the rescue of disease causative variants, the investigators will perform a stable correction of genetic variants identified through CRISPR/Cas9 gene editing approach, in u-RPC isolated from patients carrying pathogenic variants.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Meyer Children's Hospital IRCCS, Florence
  - USL Toscana Centro, Florence
  - Azienda Ospedaliero Universitaria Pisana, Pisa

IPD SHARING:
Plan to Share IPD: No